CLINICAL TRIAL: NCT03209011
Title: The Changes of CD4+T Cells Frequency and Function During Pegylated Interferon α-2a and Nucleoside Analogues Treatment in Patients With Chronic Hepatitis B
Brief Title: The Changes of CD4+T Cells Frequency and Function During Antiviral Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yao Xie (Other)
Responsible Party: Sponsor-Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Organization: Beijing Ditan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DTXY013
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B Infection
Keywords: chronic hepatitis B; hepatitis B virus; CD4+T Cells; Pegylated Interferon α-2a; Nucleoside Analogues
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): patients who were untreated ever in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly till 48 weeks.
  Interventions: Drug: Peginterferon Alfa-2a
- control group (No Intervention): patients who were untreated ever in immune-active phase took Nucleoside Analogues for maintenance treatment.

INTERVENTIONS:
Drug: Peginterferon Alfa-2a — patients untreated in immune-active phase were given subcutaneous injection of Peginterferon Alfa-2a with starting dose of 180 mg/weekly in experiment group.
  Other Names: Peg-IFN-α
  Arms: experimental group

SUMMARY:
Pegylated interferon α-2a(Peg-IFN-α) not only inhibit viral replication, but also play an important role in immune regulation, while Nucleoside analog(ue) drugs only inhibit viral replication. In hepatitis B infection, CD4+T Cells are the main effector cells in adaptive immune response. This study was aimed at investigating the changes of CD4+T Cells frequency and function, and the expression of costimulatory molecules during Peg-IFN-αand nucleoside analog(ue) therapy.Meanwhile, the investigators want to verify whether Peg IFN - alpha suppressed the virus and the reduction of virus led to the recovery of CD4+T Cells function, or Peg IFN - alpha enhanced CD4+T Cells function which gave rise to the decline of the virus.

DETAILED DESCRIPTION:
Pegylated interferon α-2a(Peg-IFN-α)and Nucleoside analog(ue) drugs can inhibit viral replication , but Peg-IFN-α also play an important role in immune regulation . In hepatitis B infection, CD4+T Cells are the main effector cells in adaptive immune response.Peg-IFN-α recommended as the first-line treatment has a higher chance to achieve HBeAg seroconversion and even HBsAg disappearance than nucleoside analog(ue) drugs, which may be related to the functional activation of CD4+T Cells in the case of hepatitis and the function enhancement of CD4+T Cells during Peg-IFN-α therapy. This study was aimed at investigating the changes of CD4+T Cells frequency and function, and the expression of costimulatory molecules during Peg-IFN-αand nucleoside analog(ue) therapy.Meanwhile, the investigators want to explore whether the decline of HBsAg and HBeAg resulted in recovery of CD4+T cells function, or recovery of CD4+T Cells function led to the decrease of HBsAg and HBeAg. Several studies demonstrated that HBsAg and HBeAg could damage CD4+T cells function, and the loss of HBsAg and HBeAg led to recovery of CD4+T cells function.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg and HBeAg positive for more than 6 months, HBV DNA detectable with ALT level abnormal lasted for three months and at least time190 IU/L or liver puncture biopsy demonstrated apparent inflammation, never treated before enrolled.

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the changes of CD4+T Cells | at baseline and at treatment week 12, 24.
  the changes of CD4+T cells%, CD62L+T cells%, CD62L-T cells%, CD62L+/ CD62L-, CD69+CD4+T cells%, CD69MFI, CD69ABC, IFN-AR2+CD4+T cells%, IFNAR2MFI, IFNAR2ABC will be measured by flow cytometry during Pegylated Interferon α-2a and Nucleoside Analogues treatment every 3 months.

SECONDARY OUTCOMES:
the change of HBVDNA levels (IU/ML) | at baseline and at treatment 12, 24, 36, 48 weeks
  the curative effect of antiviral therapy will be evaluated by HBV markers
the change of ALT levels(U/L) | at baseline and at treatment 12, 24, 36, 48 weeks
  the curative effect of antiviral therapy will be evaluated by ALT levels
the change of AST levels(U/L) | at baseline and at treatment 12, 24, 36, 48 weeks
  the curative effect of antiviral therapy will be evaluated by AST levels

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China